CLINICAL TRIAL: NCT02012348
Title: Analysis of the Effect of Antimicrobial Soap on Bacterial Survival
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Principal Investigator, Richard Gallo, Chair, Division of Dermatology, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UCSD 121622
Record Dates: First submitted 2013-12-10; First posted 2013-12-16 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Survival of Bacteria on Skin After Using Different Soaps
Keywords: bacteria survival, surfactants
MeSH Terms: interventions — triclocarban; Benzalkonium Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control soap (Placebo Comparator): Forearms of subjects in this arm will be washed with control (non-antibacterial) soap
  Interventions: Other: Control soap
- Antibacterial soap with triclocarban (Experimental): The forearms of subjects in this group will be washed with antibacterial soap containing triclocarban
  Interventions: Other: Antibacterial soap with triclocarban
- Antibacterial soap + benzalkonium chloride (Active Comparator): The forearms of subjects in this group will be washed with antibacterial soap containing benzalkonium chloride
  Interventions: Other: Antibacterial soap + benzalkonium chloride

INTERVENTIONS:
Other: Antibacterial soap with triclocarban
  Arms: Antibacterial soap with triclocarban
Other: Antibacterial soap + benzalkonium chloride
  Arms: Antibacterial soap + benzalkonium chloride
Other: Control soap
  Arms: Control soap

SUMMARY:
This study will recruit up to 10 healthy volunteers. An avirulent strain of S. pyogenes will be applied to their forearms after washing each of their forearms with different types of soap, one with an antimicrobial compound, and the other without an antimicrobial compound. After several hours of incubation, the subject's forearms will be swabbed for bacteria. The forearms will then be cleansed with antibacterial soap and water followed by 70% ethanol. The bacterial swabs will be analyzed and compared between the different soaps that were used to cleanse each digit prior to the application of S. pyogenes. The investigator expects the number of bacteria surviving on the skin of forearms washed with antimicrobial soaps will be fewer than with control soap.

DETAILED DESCRIPTION:
The study timeline will be as follows:

Day -7 to -1 - After obtaining informed consent, potential participants will be screened. A brief history and physical exam will be done on those who meet enrollment criteria. They will be assigned a start date to coincide with Day 0 below.

Day 0 - Participants will be instructed not to shower on this day. They may shower the evening before Day 0, however starting at midnight on Day 0, the participant will be advised not to shower. They will also be asked to wear a shirt with long sleeves. Significant exercise, sunbathing, and the use of creams or lotions on the forearms should also be avoided starting on Day 0, and these restrictions will remain in place until all Day 1 study-related procedures are completed. In the late afternoon on this day, the subject will have six (6) 2 cm x 2 cm squares drawn on each forearm using a skin marker. The volar forearms will be washed with soap, taking care to not remove the skin markings. One forearm will be washed with a soap containing an antibacterial compound. The other forearm will be washed using a control soap that does not contain an antibacterial compound. Each washing will consist of the application of 1.5 mL of test product to the volar forearm. A lather will be generated for 20 seconds using a gloved hand. The forearm will be rinsed with running tap water for 30 seconds and allowed to air-dry. Each forearm will be wrapped in gauze once dry. The gauze should be kept dry and in place until removed by the study staff the following day.

Day 1 - On the morning of Day 1, the gauze will be removed from participants' forearms, and 10 µL PBS containing 104 CFU of avirulent Streptococcus pyogenes (strain NZ131 M49) will be applied to the center of each of the squares previously drawn on participants' forearms. The bacteria will be spread within each square to evenly coat the surface of the skin within the square. The bacteria will then be allowed to air dry. Once dry, skin swabs will be rubbed over two of the squares on each forearm to collect a sample of the bacteria on the forearm at that location. After swabbing, these areas will be immediately disinfected with 70% alcohol. The forearms will then be wrapped again in gauze. One hour later, the gauze will be removed, and two more squares on each forearm will be swabbed for bacteria. These squares will then be disinfected with 70% alcohol, and gauze reapplied to the forearms. One hour later (two hours post-washing), the gauze will be removed, and the remaining two squares on each forearm will be swabbed for bacteria. Both forearms will then be washed with 70% ethanol and rinsed with water to remove any remaining bacteria. This will conclude the study-related procedures for Day 1. Participants are then free to shower, sunbathe, exercise and apply any creams or lotions to their forearms until the following week.

These same study procedures as above will be repeated again on Days 7 and 8, however the antibacterial soap will be used to wash one of the forearms will be replaced by a different antibacterial soap. The exact details are described in the paragraphs below.

Day 7 - Participants will be instructed not to shower on this day. They may shower the evening before Day 7, however starting at midnight on Day 7, the participant will be advised not to shower. They will also be asked to wear a shirt with long sleeves. Significant exercise, sunbathing, and the use of creams or lotions on the forearms should also be avoided starting on Day 7, and these restrictions will continue until all Day 8 study-related procedures are completed. In the late afternoon on this day, the subject will have six (6) 2 cm x 2 cm squares drawn on each forearm using a skin marker. The volar forearms will be washed with soap, taking care to not remove the skin markings. One forearm will be washed with a soap containing an antibacterial compound. The other forearm will be washed using a control soap that does not contain an antibacterial compound. Each washing will consist of the application of 1.5 mL of test product to the volar forearm. A lather will be generated for 20 seconds using a gloved hand. The forearm will be rinsed with running tap water for 30 seconds and allowed to air-dry. Each forearm will be wrapped in gauze once dry. The gauze should be kept dry and in place until removed by the study staff the following day.

Day 8 - On the morning of Day 8, the gauze will be removed from participants' forearms, and 10 µL PBS containing 104 CFU of avirulent Streptococcus pyogenes (strain NZ131 M49) will be applied to the center of each of the squares previously drawn on participants' forearms. The bacteria will be spread within each square to evenly coat the surface of the skin within the square. The bacteria will then be allowed to air dry. Once dry, skin swabs will be rubbed over two of the squares on each forearm to collect a sample of the bacteria on the forearm at that location. After swabbing, these areas will be immediately disinfected with 70% alcohol. The forearms will then be wrapped again in gauze. One hour later, the gauze will be removed, and two more squares on each forearm will be swabbed for bacteria. These squares will then be disinfected with 70 alcohol, and gauze reapplied to the forearms. One hour later (two hours post-washing), the gauze will be removed, and the remaining two squares on each forearm will be swabbed for bacteria. Both forearms will then be washed with 70% ethanol and rinsed with water to remove any remaining bacteria. This will conclude all study-related procedures. Participants are then free to shower, sunbathe, exercise and apply any creams or lotions to their forearms.

ELIGIBILITY:
Inclusion Criteria:

Those who meet all of the following criteria are eligible for enrollment into the study:

1. Age 18-60 years
2. Male or female of any race and ethnicity
3. Subject agrees to comply with study requirements.

Exclusion Criteria:

1. Subjects with severe medical condition(s) that in the view of the investigator prohibits participation in the study
2. Dermatologic disease such as psoriasis or atopic dermatitis which may have inherently abnormal antimicrobial peptide levels
3. Subject has Netherton's syndrome or other genodermatoses that result in a defective epidermal barrier
4. Pregnant or nursing females
5. Immunocompromised subjects (e.g., lymphoma, HIV/AIDS, Wiskott-Aldrich Syndrome), or with a history of active or malignant disease (excluding non-melanoma skin cancer) as determined by the participant's medical history.
6. Subjects with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol
7. Subjects with significant concurrent medical condition(s) at screening that in the view of the investigator prohibits participation in the study (e.g., severe concurrent allergic disease, condition associated with malignancy, and condition associated with immunosuppression)
8. Active viral or fungal skin infections at the target areas
9. Are currently receiving lithium, antimalarials, or intramuscular gold now or within the last 4 weeks.
10. Ongoing participation in an investigational drug trial
11. Use of any oral or topical antibiotic during the study and up to one week prior to entering the study
12. Use of any local topical medications less than one week prior to screening
13. Use of any systemic immunosuppressive therapy less than four weeks prior to screening.
14. Subjects with a history of or propensity to developing reactions after use of over the counter cleansers
15. Subjects with diabetes
16. Injured, broken skin that, per the investigator, may cause injury if exposed to low virulence GAS.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Dermatology, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Soap: Forearms of subjects in this arm will be washed with control (non-antibacterial) soap
  Control soap
- Antibacterial Soap With Triclocarban: The forearms of subjects in this group will be washed with antibacterial soap containing triclocarban
  Antibacterial soap with triclocarban
- Antibacterial Soap + Benzalkonium Chloride: The forearms of subjects in this group will be washed with antibacterial soap containing benzalkonium chloride
  Antibacterial soap + benzalkonium chloride
Period: Overall Study
Arm/Group | Control Soap | Antibacterial Soap With Triclocarban | Antibacterial Soap + Benzalkonium Chloride
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Soap | Antibacterial Soap With Triclocarban | Antibacterial Soap + Benzalkonium Chloride | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (5) | 32.2 (5) | 32.2 (5) | 32.2 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 12
  Male | 6 | 6 | 6 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 3 | 3 | 3 | 9
  Unknown or Not Reported | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Relative GAS Survival
Description: A skin swab will be used to measure the bacterial survival 30 minutes after bacteria application and soap treatment. The bacteria being applied and subsequently measured is Group A Streptococcus (GAS). The bacterial survival is expressed as abundance of GAS relative to abundance of other bacterial species isolated from the swab.
Time Frame: 30 minutes post-bacteria application
Measure: Mean (Standard Error); unit: percentage overall bacterial abundance
Arm/Group | Control Soap | Antibacterial Soap With Triclocarban | Antibacterial Soap + Benzalkonium Chloride
Number analyzed (Participants) | 10 | 10 | 10
percentage overall bacterial abundance | 100 (15) | 75 (20) | 90 (21.7)

2. Secondary Outcome: Relative GAS Survival
Description: A skin swab will be used to measure the bacterial survival 1 hour after bacteria application (2 hours post washing with soap). The bacteria being applied and subsequently measured is Group A Streptococcus (GAS). The bacterial survival is expressed as abundance of GAS relative to abundance of other bacterial species isolated from the swab.
Time Frame: 1 hour after bacteria application / 2 hours post washing
Measure: Mean (Standard Error); unit: percentage overall bacterial abundance
Arm/Group | Control Soap | Antibacterial Soap With Triclocarban | Antibacterial Soap + Benzalkonium Chloride
Number analyzed (Participants) | 10 | 10 | 10
percentage overall bacterial abundance | 100 (12.5) | 86.7 (23.3) | 61.7 (13.3)

ADVERSE EVENTS:
Arm/Group | Control Soap | Antibacterial Soap With Triclocarban | Antibacterial Soap + Benzalkonium Chloride
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No